CLINICAL TRIAL: NCT02049151
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Trial of Tecemotide Versus Placebo in Subjects With Completed Concurrent Chemo-radiotherapy for Unresectable Stage III Non-small Cell Lung Cancer (NSCLC)
Brief Title: Tecemotide Following Concurrent Chemo-radiotherapy for Non-small Cell Lung Cancer
Acronym: START2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is terminated prematurely as the sponsor decided to discontinue program with Tecemotide in NSCLC
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR 63325-021; 2013-003760-30 (EudraCT Number)
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Tecemotide; Placebo; NSCLC; L-BLP25
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — L-BLP25; Cyclophosphamide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tecemotide (Experimental)
  Interventions: Drug: Tecemotide; Drug: Cyclophosphamide (CPA)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Saline (sodium chloride)

INTERVENTIONS:
Drug: Tecemotide — Tecemotide injection will be administered once weekly subcutaneously at a dose of 806 microgram up to Week 8 and from Week 14, every 6 weeks until end-of-trial, or until NSCLC progression.
  Arms: Tecemotide
Drug: Placebo — Matching placebo injection will be administered once weekly subcutaneously up to Week 8 and from Week 14, every 6 weeks until end-of-trial, or until NSCLC progression.
  Arms: Placebo
Drug: Cyclophosphamide (CPA) — CPA injection will be administered as a single intravenous infusion at a dose of 300 milligram per square meter (mg/m^2) (to a maximum of 600 mg) 3 days before the first injection of tecemotide.
  Arms: Tecemotide
Drug: Saline (sodium chloride) — Matching placebo (saline) injection will be administered as a single intravenous (0.9 percent [%] sodium chloride) infusion 3 days before the first injection of tecemotide-matching placebo.
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, placebo-controlled, randomized, Phase 3 trial in subjects with unresectable stage III non-small cell lung cancer (NSCLC) who have demonstrated either stable disease or objective response following primary concurrent chemo-radiotherapy (CRT), comparing overall survival (OS) time in subjects treated with tecemotide versus subjects treated with tecemotide-matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, before any trial-related activities are carried out
* Histologically or cytologically documented unresectable stage III NSCLC, including bronchioalveolar carcinomas. Cancer stage must be confirmed and documented by computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET) scan
* Prior concurrent CRT which is defined as follows:

  * Minimum of 2 cycles of platinum-based chemotherapy
  * Radiotherapy with a total tumor dose greater than equal to (>=) 60 Gray and a single fraction dose >= 1.8 Gray
  * Overlap of radiotherapy with minimum 2 cycles of platinum-based chemotherapy (one cycle is defined as either 3 or 4 weeks depending on the chemotherapy regimen). A deviation of 2 to 3 days from an exact overlap is acceptable. Purely radiosensitizing doses of chemotherapy are not acceptable (for example [e.g.], daily low dose regimens; weekly carbo-platinum + paclitaxel regimens are allowed).
* Subjects must have completed the primary thoracic CRT at least 4 weeks (28 days) and no later than 12 weeks (84 days) prior to randomization. Subjects who received prophylactic brain irradiation as part of primary CRT are eligible.
* Documented stable disease or objective response, according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, after primary concurrent CRT for unresectable stage III disease, within 4 weeks (28 days) prior to randomization
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* A platelet count, white blood cells (WBC) and hemoglobin value as defined in the protocol
* Male or female, greater than or equal to 18 years of age
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Undergone lung cancer specific therapy (including surgery) other than initial concurrent CRT
* Received chemotherapy during radiotherapy in radiosensitizing doses only (e.g., daily low dose regimens; weekly carbo-platinum + paclitaxel regimens are allowed).
* Metastatic disease
* Malignant pleural effusion at initial diagnosis, during initial CRT, and/or at trial entry
* Past or current history of neoplasm other than lung carcinoma, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years
* A recognized immunodeficiency disease including human immunodeficiency virus (HIV) infection and other cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have hereditary, congenital or acquired immunodeficiencies
* Splenectomy
* Any preexisting medical condition requiring chronic systemic steroid or immunosuppressive therapy (steroids for the treatment of radiation pneumonitis are allowed)
* Receipt of immunotherapy (as defined in the protocol) within 4 weeks prior to randomization
* Receipt of investigational systemic drugs (including off-label use of approved products) within 4 weeks prior to randomization
* Autoimmune disease
* Active or chronic infectious hepatitis
* Infectious process that, in the opinion of the Investigator, could compromise the subject's ability to mount an immune response
* Clinically significant hepatic dysfunction, renal dysfunction and cardiac disease as defined in the protocol
* Pregnant or breast-feeding women
* Known drug abuse/alcohol abuse
* Participation in another interventional clinical trial within the past 28 days (excluding purely observational studies)
* Requires concurrent treatment with a non-permitted drug
* Known hypersensitivity to any of the trial treatment ingredients
* Legal incapacity or limited legal capacity
* Any other reason that, in the opinion of the Investigator, precludes the subject from participating in the trial
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (2):
- Please Contact U.S. Medical Information Located in, Rockland, Massachusetts, United States
- Please contact the Merck KGaA Communication Center Located in, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject(informed consent): 21 Mar 2014/11 Sep 2014. Study completion date: 02 Jul 2015.
Pre-assignment Details: 50 subjects were screened for eligibility; 15 excluded (mainly due to non-fulfillment of inclusion or exclusion criteria) and 35 subjects were randomized. Three subjects were randomized but were not treated.
Groups:
- Tecemotide (L-BLP25) + Cyclophosphamide: Single dose of cyclophosphamide (300 milligrams per square meter [mg/m^2] to a maximum of 600 mg) was administered intravenously, 3 days prior to the tecemotide dosing, tecemotide (L-BLP25) (806 micrograms [mcg]) was administered weekly subcutaneously for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with tecemotide (L-BLP25) (806 mcg) were administered every 6 weeks until disease progression was documented.
- Placebo + Saline: Single dose of saline (sodium chloride, 9 grams per liter [g/L]) was administered intravenously, 3 days prior to the tecemotide dosing, placebo doses matched to tecemotide (L-BLP25) was administered weekly subcutaneously for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with placebo were administered every 6 weeks until disease progression was documented.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Started | 15 (2 subjects did not receive treatment) | 17 (1 subject did not receive treatment)
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all subjects who had taken at least one dose of trial treatment (tecemotide [L-BLP25] or placebo), including cyclophosphamide or saline.
Groups:
- Tecemotide (L-BLP25) + Cyclophosphamide: Single dose of cyclophosphamide (300 mg/m^2 to a maximum of 600 mg) was administered intravenously, 3 days prior to the tecemotide dosing, tecemotide (L-BLP25) (806 mcg) was administered weekly subcutaneously for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with tecemotide (L-BLP25) (806 mcg) were administered every 6 weeks until disease progression was documented.
- Placebo + Saline: Single dose of saline (sodium chloride, 9 g/L) was administered intravenously, 3 days prior to the tecemotide dosing, placebo doses matched to tecemotide (L-BLP25) was administered weekly subcutaneously for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with placebo were administered every 6 weeks until disease progression was documented.
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline | Total Title
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age Continuous | 66.2 (5.99) | 63.9 (10.45) | 65.0 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time (in months) from randomization to death. Data has been presented in terms of number subjects who died and number of censored subjects.
Time Frame: Time from date of randomization until death, assessed maximum up to 16 months
Population: Safety Analysis Set included all subjects who had taken at least one dose of trial treatment (tecemotide [L-BLP25] or placebo), including cyclophosphamide or saline. Analysis was not performed due to the premature termination of this study and the tecemotide program based on negative results in EMR 63325-009 (NCT00960115).
Measure: Number; unit: subjects
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 15 | 17
subjects
  Number of deaths | 1 | 2
  Number for censored | 14 | 15

2. Secondary Outcome: Time to Symptom Progression (TTSP)
Description: TTSP was measured from date of randomization to date of disease progression (defined based on RECIST v1.1), using the lung cancer symptom scale (LCSS), a validated questionnaire consisting of an observer scale and a subject scale used to specifically measure symptom changes relevant to quality of life (QoL) for individuals undergoing treatment for lung cancer. Subject scale was used as a tool to determine TTSP. It was a 9-item questionnaire used to document subject-reported outcomes for a variety of lung cancer associated symptoms. The average symptomatic burden index (ASBI) was used to determine differences in the treatment groups. ASBI was the mean of the 6 symptom scores derived from the LCSS questionnaire. Symptom progression was defined as an increase (worsening) of the ASBI score of 10% of the scale breadth (10 mm on a scale of 0-100 mm) from the baseline score on at least 2 consecutive assessments during the period when assessments are performed every 3 weeks and every 6 weeks.
Time Frame: Time from date of randomization until progressive disease (PD), assessed up to 16 months
Population: Analysis was not performed due to the premature termination of this study and the tecemotide program based on negative results in EMR 63325-009 (NCT00960115).
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from date of randomization until date of the first documentation of PD or death due to any cause in the absence of documented PD, whichever occurred first. PFS was assessed as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). PD was defined as at least a 20% increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Subjects without event were censored on the date of last tumor assessment.
Time Frame: Time from date of randomization until PD or death, assessed up to 16 months
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP was measured from the date of randomization to the date of tumor progression. Date of tumor progression was date of radiological diagnosis of PD, performed as per RECIST 1.1. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression. For participants alive without tumor progression at time of analysis, the time between date of randomization and date of last trial treatment was calculated and used as a censored observation in the analysis. Subjects dying from causes other than PD was censored at time of death.
Time Frame: Time from date of randomization until PD, assessed up to 16 months
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, National Cancer Institute-Common Toxicity Criteria (NCI-CTC)Grade 3/4 TEAEs, TEAEs Leading to Permanent Discontinuation, TEAEs Leading to Death, Injection Site Reactions (ISRs)
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs occurred between the first dose of study drug and up to 42 days after the last dose that were absent before treatment or that worsened relative to pretreatment state. Number of Subjects With TEAEs, Serious TEAEs, NCI-CTC Grade 3/4 TEAEs, TEAEs Leading to Permanent Discontinuation, TEAEs Leading to Death, and ISRs were reported.
Time Frame: Time from first dose up to 42 days after the last dose of the trial treatment: assessed maximum up to 16 months
Population: as for baseline characteristics
Measure: Number; unit: subjects
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 15 | 17
subjects
  TEAEs | 14 | 13
  Serious TEAEs | 4 | 1
  Grade 3 or 4 TEAEs | 5 | 2
  TEAEs Leading to Permanent Discontinuation | 2 | 1
  TEAEs leading to death | 0 | 0
  ISRs | 0 | 3

ADVERSE EVENTS:
Time Frame: Time from first dosing day until 42 days following the last vaccination of tecemotide (L-BLP25) or placebo assessed maximum up to 16 months.
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Serious Adverse Events (participants affected / at risk) | 4/15 | 1/17
Other Adverse Events (participants affected / at risk) | 14/15 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) + Cyclophosphamide (N=15) | Placebo + Saline (N=17)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) + Cyclophosphamide (N=15) | Placebo + Saline (N=17)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 3
Feeling hot (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 1
Injection site hypoaesthesia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 2
Lethargy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Sponsor discontinued development of tecemotide (L-BLP25) in NSCLC, hence the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication will be publication of results of the analysis of primary endpoint(s) that will include data from all trial centers. Any publications and presentations of results, either in whole or in part, by investigators or their representatives will require pre-submission review by the sponsor/CRO. Sponsor will not suppress or veto publications, but maintains right to delay publication in order to protect intellectual property rights.